CLINICAL TRIAL: NCT02930720
Title: The Influence of Various Breathing Protocols and Cough on the Amount of Pelvic Floor Displacement in Women With Stress Urinary Incontinence and Healthy Women: An Ultrasound Study
Brief Title: Pelvic Floor Displacement in Women With SUI and Healthy Women: An Ultrasound Study (Stress Urinary Incontinence)
Acronym: SUI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assuta Hospital Systems (Other)
Responsible Party: Principal Investigator, Iris sinai, Director, Assuta Hospital Systems
Other Study IDs: AssutaHS0087-16
Record Dates: First submitted 2016-10-10; First posted 2016-10-12 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Healthy; Stress Urinary Incontinence
Keywords: TAUS; breathing protocols and cough; pelvic floor displacement; women; SUI
MeSH Terms: conditions — Urinary Incontinence, Stress; Cough

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Pelvic floor main role is to maintain continence. pelvic floor malfunction could lead to urinary incontinence (UI). The known prevalence of UI among women is 25%-72%, in about 25%-50% it is Stress Urinary Incontinence (SUI), SUI prevalence changes with age and obstetric history. SUI is the complaint of involuntary leakage on activities which involves inter abdominal pressure rase, such as effort or exertion, or sneezing or coughing. pelvic floor movement is coordinated with the diaphragm, it moves caudally while inhaling and cranially while exhaling. it was shown that cranial sagittal displacement of the pelvic floor is correlated to pelvic floor normal and efficient function. in order to maintain continence while internal abdominal pressure rises the pelvic floor as to work in a precise trajectory, timing and force. observing the Urinary bladder by trans abdominal ultra sound (TAUS) was found as a valid and reliable way to estimate pelvic floor sagittal displacement and function.

DETAILED DESCRIPTION:
50 women between the age 25-50 with a history of one vaginal delivery will be recruited for the study. 25 women who complain about stress urinary incontinence (research group) and 25 healthy women (control group). all research participants will sign first a participant consent form. all participants will be interviewed about their own delivery, measured for weight and height and follow a trans abdominal ultra sound (TAUS) examination. the research group participants will be asked to fill a quality of life questionaire concerning their SUI complaint.

at the TAUS examination the participant will be asked to perform:

1. 3 times quiet breathing.
2. 3 times forced exhalation.
3. 3 times cough. while doing so an ultra sound image of the urinary bladder will be saved for displacement measurements.

ELIGIBILITY:
Inclusion Criteria:

* women after one vaginal delivery on term.
* women aged 25-50
* members of 'macabi medical services'

Exclusion Criteria:

* pregnancy
* nulliparous women
* women who had C section delivery
* known neurologic disease
* previous history of pelvic or back surgery
* previous history of pelvic fracture
* known pulmonary disease
* active urinary tract infection

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 50 parous women, who performed one vaginal delivey. age 25-50. all women are 'macabi medical services' members. 25 women who complain about stress urinary incontinence. 25 healthy women.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-08 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
pelvic floor displacement | 20-30 minutes
  in mm

SECONDARY OUTCOMES:
Incontinence Quality of Life (I-QOL) | 5 minutes
  score of questionaire

CONTACTS AND LOCATIONS:
Locations (1):
- Macabi hadar yossef, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No